CLINICAL TRIAL: NCT05133648
Title: Association of Anesthesia Technique With Morbidity and Mortality in Patients With COVID-19 and Surgery for Hip Fracture: a Retrospective Population Cohort Study
Brief Title: Anesthesia Technique in COVID-19 Positive Hip Fracture Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Janny Ke, Clinical Assistant Professor, University of British Columbia
Other Study IDs: H22-03212
Record Dates: First submitted 2021-11-21; First posted 2021-11-24 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Hip Fractures; COVID-19; General Anesthesia; Spinal Anesthesia
MeSH Terms: conditions — Hip Fractures; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hip Surgery without COVID-19 infection: January to December 2021
  Interventions: Procedure: Hip Fracture Surgery
- Hip Surgery with COVID-19 infection: January to December 2021
  Interventions: Procedure: Hip Fracture Surgery; Other: COVID-19 infection
- Hip Surgery pre-pandemic: January 2017 to December 2019
  Interventions: Procedure: Hip Fracture Surgery

INTERVENTIONS:
Procedure: Hip Fracture Surgery — Hip fracture surgery
Other: COVID-19 infection — COVID-19 infection
  Groups: Hip Surgery with COVID-19 infection

SUMMARY:
Patients with COVID undergoing hip fracture repair have high mortality rates. If spinal anesthesia is associated with decreased rates of mortality, this study could provide hypothesis generating data for prospective studies. Investigators hypothesize that spinal anesthesia (SA) is associated with decreased mortality compared to general anesthesia (GA) for patients undergoing hip fracture surgery. The primary objective is to determine for patients undergoing hip surgery with COVID-19 infection, whether SA, as compared to GA, is associated with a lower rate of mortality 30 days postoperatively. The secondary objective is to determine whether SA, as compared to GA, is associated with a lower rate of morbidity 30 days postoperatively. Investigators will be analyzing a data set provided by the National Surgical Quality Improvement Program (NSQIP). Descriptive statistics will be performed. Multivariable logistic regression will be performed for the primary and secondary objectives.

DETAILED DESCRIPTION:
Background: Patients with hip fracture have poor outcomes, attributed to risk factors that include advanced age and higher rates of underlying chronic comorbidities. COVID-19 infection is an independent risk factor for increased mortality in hip fracture patients in the perioperative period. A recent meta-analysis demonstrates COVID-19 infection is associated with higher than seven-fold increase in risk of mortality. Recommended management of hip fracture includes timely surgical repair, multimodal pain control, and multidisciplinary follow-up, to facilitate return to mobility and independent function.

Anesthesia for hip fracture surgery can be achieved by either general anesthesia (GA) or spinal anesthesia (SA). The potential advantages of SA include opioid-sparing effects, lessened impacts on the respiratory and gastrointestinal systems, and reduction in rates of adverse outcomes such as pneumonia, mechanical ventilation, intensive care unit (ICU) admission, venous thromboembolism (VTE), myocardial infarction (MI), stroke, transfusion, readmission, and prolonged postoperative length of stay. However, a recent randomized control trial found no difference between SA and GA for older adults undergoing hip fracture surgery for the primary outcome of survival and recovery of ambulation at 60 days.

While emerging evidence shows COVID-19 infection increases mortality after hip surgery, there is a lack of research examining whether the choice of anesthetic technique modifies the postoperative mortality and morbidity of hip fracture patients with COVID-19 infection. This is particularly important due to the high mortality (35% in COVID-positive patients, vs. 2% in patients without COVID), with the potential for SA to modify this risk by circumventing the need for airway interventions. SA may also offer superiority over general anesthesia for limiting aerosol generation and exposure of operating room staff during the pandemic. While SA may reduce the risk of pulmonary morbidity by reducing the need for airway interventions, its motor block on accessory muscles and the need for sedation may adversely impact ventilation. Investigators hypothesize that spinal anesthesia (SA) is associated with decreased mortality compared to general anesthesia (GA) for patients undergoing hip fracture surgery.

Study Design: The requirement for written informed consent will be waived for use of deidentified data. Patient information will be obtained for the retrospective cohort analysis using the NSQIP® (general dataset linked with the Hip Fracture Procedure Targeted Dataset), a prospectively-collected multicentre dataset with more than 150 clinical variables within 30 days after surgery. The setting of this study will be patient data obtained from the multicentre generated NSQIP Hip Fracture Procedure Targeted Dataset. The period of patient data obtained will include from January 2017 through December 2021. We will omit the data from January 2020 to December 2020 given there was no reporting of COVID status during this period. Data will only be obtained from patients undergoing hip surgery with mortality and morbidity gathered for 30 days postoperatively. In this study, the investigators goal is to evaluate the adjusted association between anesthesia technique and mortality and morbidity after hip fracture surgery for patients who tested positive for COVID-19.

The primary objective is to determine for patients undergoing hip surgery with COVID-19 infection, whether SA, as compared to GA, is associated with a lower rate of mortality 30 days postoperatively.

Our secondary objective is to determine whether SA, as compared to GA, is associated with a lower rate of morbidity 30 days postoperatively. To provide context for interpretation, we will describe the epidemiology of the following rates during versus before the 2020 COVID-19 pandemic (January to December 2021, compared to 2017 to 2019): 1) SA versus GA uti-lization for hip fracture surgery, and 2) mortality and morbidity for hip surgery patients without COVID-19 infection. Finally, we will quantify the mortality and morbidity for pa-tients with versus without COVID-19 infection undergoing hip fracture surgery, stratified by SA and GA.

Purpose: The purpose of this study is to evaluate the adjusted association between anesthesia technique and mortality and morbidity after hip fracture surgery

Population cohorts: The study will be divided into three cohorts: those undergoing hip surgery 1) without COVID-19 infection January to December 2021, 2) with COVID-19 infection January to December 2021, and 3) pre-pandemic from January 2017 to December 2019.

Due to the variable duration of asymptomatic period that can precede symptoms and diagnosis, COVID-19 infection status will be classified as follows.

In the primary analysis, COVID-negative patients will be defined as no preoperative COVID (within 14 days before surgery) and no postoperative COVID, and COVID-positive patients will be defined as yes (lab-confirmed) preoperative COVID and no postoperative COVID. In NSQIP, preoperative COVID status denotes within 14 days be-fore surgery, and patients with preoperative COVID are always coded "No" for postopera-tive COVID. NSQIP does not have previous history of COVID prior to 14 days, which is a major limitation given the increased mortality of patients with recent COVID undergoing surgery (24).

In NSQIP, preoperative COVID status denotes within 14 days before surgery, and patients with preoperative COVID are always coded "No" for postoperative COVID. NSQIP does not have previous history of COVID prior to 14 days, which is a major limitation given the increased mortality of patients with recent COVID undergoing surgery.

As patients with postoperative COVID-positive status are difficult to interpret due to variable incubation period and the possibility of COVID-19 contraction while in hospital postoperatively, investigators will perform sensitivity analysis using alternative definitions for the COVID-positive cohort, including 1) laboratory confirmed preoperatively or postoperatively, 2) laboratory confirmed or symptomatic preoperatively, and 3) suspected and laboratory confirmed anytime preoperatively or postoperatively).

Data analysis: Investigators will be analyzing a data set provided by the National Surgical Quality Improvement Program (NSQIP). Descriptive statistics will be performed. Multivariable logistic regression will be performed for the primary and secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Sampled in the NSQIP Hip Fracture Procedure Targeted Dataset from January 2017 through December 2019 and from January 2021 to December 2021.
* undergoing surgical fixation of hip fractures using either general and/or spinal anesthesia.
* In case of reduced Procedure-Targeted data collection during the COVID-19 pandemic, investigators will also create a total open hip fracture cohort using relevant Current Procedural Terminology codes (27244, 27245, 27269, 27236, or 27248)

Exclusion Criteria:

* Primary or secondary anesthetic technique listed as local anesthesia alone, local anesthesia with intravenous sedation, epidural, and those with no reported anesthesia technique
* American Society of Anesthesiologists (ASA) Physical Status (PS) V (defined as "5-Moribund"), and
* Ventilator-dependence preoperatively.
* Platelet counts less than 80,000/mm3 within 90 days before surgery,
* International normalized ratio (INR) greater than or equal to 1.5, or
* Partial thromboplastin time (PTT) greater than 35 seconds (likelihood of being ineligible for SA)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include all patients 19 years or older who are sampled in the NSQIP Hip Fracture Procedure Targeted Dataset from January 2017 through December 2019 and January 2021 to December 2021 undergoing surgical fixation of hip fractures using either general and/or spinal anesthesia.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-03 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days post operatively
  All-cause 30-day mortality following hip fracture surgery.

SECONDARY OUTCOMES:
Stroke or cerebrovascular accident (CVA) | Within 30 days post operatively
  Occurrence of a stroke or cerebrovascular accident (CVA) within 30 days following hip fracture surgery (Yes, or No).
Myocardial Infarction (MI) | Within 30 days post operatively
  Occurrence of a Myocardial Infarction intraoperatively or within 30 days following hip fracture surgery
Postoperative Delirium | Within 30 days post operatively
  Occurrence of postoperative delirium within 30 days following hip fracture surgery (Yes, or No).
Pneumonia | Within 30 days post operatively
  Occurrence of pneumonia within 30 days following hip fracture surgery (Yes, or No).
Acute Renal Failure | Within 30 days post operatively
  Occurrence of acute renal failure up to 30 days following hip fracture surgery (Yes, or No).
Transfusion | Within 30 days post operatively
  Participant had bleeding requiring a transfusion within 30 days following hip fracture surgery (Yes, or No).
Post-Operative Ventilation | Within 30 days post operatively
  Participant having a total cumulative duration of ventilator-assisted respirations greater than 48 hours during the postoperative hospitalization or any other time within 30 days following hip fracture surgery (Yes, or No).
Hospital Readmission | Within 30 days post operatively
  Participant readmitted to hospital within 30 days following hip fracture surgery (Yes, or No).
Unplanned Reoperation | Within 30 days post operatively
  Occurrence of an unplanned reoperation within 30 days following hip fracture surgery (Yes, or No).
Length of Stay | Post-operative period in hospital, on average 5 days
  Total number of days from the day of operation to the day of discharge from hospital
Hospital Stay greater than 30 days | Greater than 30 days postoperatively
  If the participant has not yet been discharged from the acute care setting within 30 days after the primary procedure (Yes, or No).
Discharge Destination | Postoperative Period at Time of discharge, on average 5 days
  Destination after discharge from hospital (home or not home)
Venous Thromboembolism | Within 30 days post operatively
  Composite outcome of the occurrence of a pulmonary embolism or deep venous thrombosis within 30 days following hip fracture surgery.
Sepsis | Within 30 days post operatively
  Composite outcome of the occurrence of sepsis or septic shock within 30 days following hip fracture surgery.
Any Complication or Death | Within 30 days post operatively
  Composite outcome of the occurrence of any complication or participant deceased up to 30 days following hip fracture surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Janny Xue Chen Ke, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Hu F, Jiang C, Shen J, Tang P, Wang Y. Preoperative predictors for mortality following hip fracture surgery: a systematic review and meta-analysis. Injury. 2012 Jun;43(6):676-85. doi: 10.1016/j.injury.2011.05.017. Epub 2011 Jun 17. PMID 21683355
- [Background] Panula J, Pihlajamaki H, Mattila VM, Jaatinen P, Vahlberg T, Aarnio P, Kivela SL. Mortality and cause of death in hip fracture patients aged 65 or older: a population-based study. BMC Musculoskelet Disord. 2011 May 20;12:105. doi: 10.1186/1471-2474-12-105. PMID 21599967
- [Background] Sheikh HQ, Hossain FS, Aqil A, Akinbamijo B, Mushtaq V, Kapoor H. A Comprehensive Analysis of the Causes and Predictors of 30-Day Mortality Following Hip Fracture Surgery. Clin Orthop Surg. 2017 Mar;9(1):10-18. doi: 10.4055/cios.2017.9.1.10. Epub 2017 Feb 13. PMID 28261422
- [Background] De C, Harbham PK, Postoyalko C, Bhavanasi B, Paringe V, Theivendran K. Mortality Following Hip Fracture Surgery During COVID-19 Pandemic Compared to Pre-COVID-19 Period: A Case Matched Cohort Series. Malays Orthop J. 2021 Jul;15(2):107-114. doi: 10.5704/MOJ.2107.016. PMID 34429830
- [Background] Fell A, Malik-Tabassum K, Rickman S, Arealis G. Thirty-day mortality and reliability of Nottingham Hip Fracture Score in patients with COVID19 infection. J Orthop. 2021 Jul-Aug;26:111-114. doi: 10.1016/j.jor.2021.07.009. Epub 2021 Jul 16. PMID 34305350
- [Background] Zamora T, Sandoval F, Demandes H, Serrano J, Gonzalez J, Lira MJ, Klaber I, Carmona M, Botello E, Schweitzer D. Hip Fractures in the Elderly During the COVID-19 Pandemic: A Latin-American Perspective With a Minimum 90-Day Follow-Up. Geriatr Orthop Surg Rehabil. 2021 Jul 9;12:21514593211024509. doi: 10.1177/21514593211024509. eCollection 2021. PMID 34290897
- [Background] Cuthbert R, Ferguson D, Kayani B, Haque S, Ali A, Parkar A, Bates P, Vemulapalli K. Evidence-based approach to providing informed consent for hip fracture surgery during the COVID-19 era. World J Orthop. 2021 Jun 18;12(6):386-394. doi: 10.5312/wjo.v12.i6.386. eCollection 2021 Jun 18. PMID 34189076
- [Background] Kumar A, Haider Y, Passey J, Khan R, Gaba S, Kumar M. Mortality Predictors in Covid-19 Positive Patients with Fractures: A Systematic Review. Bull Emerg Trauma. 2021 Apr;9(2):51-59. doi: 10.30476/BEAT.2021.87742. PMID 34150914
- [Background] Grassi A, Andriolo L, Golinelli D, Tedesco D, Rosa S, Gramegna P, Ciaffi J, Meliconi R, Landini MP, Filardo G, Fantini MP, Zaffagnini S. Higher 90-Day Mortality after Surgery for Hip Fractures in Patients with COVID-19: A Case-Control Study from a Single Center in Italy. Int J Environ Res Public Health. 2021 May 13;18(10):5205. doi: 10.3390/ijerph18105205. PMID 34068405
- [Background] Balakumar B, Nandra RS, Woffenden H, Atkin B, Mahmood A, Cooper G, Cooper J, Hindle P. Mortality risk of surgically managing orthopaedic trauma during the COVID-19 pandemic. Bone Jt Open. 2021 May;2(5):330-336. doi: 10.1302/2633-1462.25.BJO-2020-0189.R1. PMID 34027674
- [Background] Alcock H, Moppett EA, Moppett IK. Early mortality outcomes of patients with fragility hip fracture and concurrent SARS-CoV-2 infection : a systematic review and meta-analysis. Bone Jt Open. 2021 May;2(5):314-322. doi: 10.1302/2633-1462.25.BJO-2020-0183.R1. PMID 34003031
- [Background] Lim MA, Pranata R. Coronavirus disease 2019 (COVID-19) markedly increased mortality in patients with hip fracture - A systematic review and meta-analysis. J Clin Orthop Trauma. 2021 Jan;12(1):187-193. doi: 10.1016/j.jcot.2020.09.015. Epub 2020 Sep 17. PMID 32958988
- [Background] Mittal R, Banerjee S. Proximal femoral fractures: Principles of management and review of literature. J Clin Orthop Trauma. 2012 Jun;3(1):15-23. doi: 10.1016/j.jcot.2012.04.001. Epub 2012 Jun 16. PMID 25983451
- [Background] Griffiths R, Babu S, Dixon P, Freeman N, Hurford D, Kelleher E, Moppett I, Ray D, Sahota O, Shields M, White S. Guideline for the management of hip fractures 2020: Guideline by the Association of Anaesthetists. Anaesthesia. 2021 Feb;76(2):225-237. doi: 10.1111/anae.15291. Epub 2020 Dec 2. PMID 33289066
- [Background] Jakobsson J, Johnson MZ. Perioperative regional anaesthesia and postoperative longer-term outcomes. F1000Res. 2016 Oct 11;5:F1000 Faculty Rev-2501. doi: 10.12688/f1000research.9100.1. eCollection 2016. PMID 27785357
- [Background] Capdevila X, Moulard S, Plasse C, Peshaud JL, Molinari N, Dadure C, Bringuier S. Effectiveness of Epidural Analgesia, Continuous Surgical Site Analgesia, and Patient-Controlled Analgesic Morphine for Postoperative Pain Management and Hyperalgesia, Rehabilitation, and Health-Related Quality of Life After Open Nephrectomy: A Prospective, Randomized, Controlled Study. Anesth Analg. 2017 Jan;124(1):336-345. doi: 10.1213/ANE.0000000000001688. PMID 27918333
- [Background] Wignall A, Giannoudis V, De C, Jimenez A, Sturdee S, Nisar S, Pandit H, Gulati A, Palan J. The impact of COVID-19 on the management and outcomes of patients with proximal femoral fractures: a multi-centre study of 580 patients. J Orthop Surg Res. 2021 Feb 24;16(1):155. doi: 10.1186/s13018-021-02301-z. PMID 33627153
- [Background] Cappelleri G, Fanelli A, Ghisi D, Russo G, Giorgi A, Torrano V, Lo Bianco G, Salomone S, Fumagalli R. The Role of Regional Anesthesia During the SARS-CoV2 Pandemic: Appraisal of Clinical, Pharmacological and Organizational Aspects. Front Pharmacol. 2021 Jun 4;12:574091. doi: 10.3389/fphar.2021.574091. eCollection 2021. PMID 34149401
- [Background] Maxwell BG, Spitz W, Porter J. Association of Increasing Use of Spinal Anesthesia in Hip Fracture Repair With Treating an Aging Patient Population. JAMA Surg. 2020 Feb 1;155(2):167-168. doi: 10.1001/jamasurg.2019.4471. PMID 31746959
- [Background] van Veen JJ, Nokes TJ, Makris M. The risk of spinal haematoma following neuraxial anaesthesia or lumbar puncture in thrombocytopenic individuals. Br J Haematol. 2010 Jan;148(1):15-25. doi: 10.1111/j.1365-2141.2009.07899.x. Epub 2009 Sep 22. PMID 19775301
- [Background] Gulur P, Tsui B, Pathak R, Koury KM, Lee H. Retrospective analysis of the incidence of epidural haematoma in patients with epidural catheters and abnormal coagulation parameters. Br J Anaesth. 2015 May;114(5):808-11. doi: 10.1093/bja/aeu461. Epub 2015 Jan 22. PMID 25614136
- [Background] Horlocker TT, Wedel DJ, Rowlingson JC, Enneking FK, Kopp SL, Benzon HT, Brown DL, Heit JA, Mulroy MF, Rosenquist RW, Tryba M, Yuan CS. Regional anesthesia in the patient receiving antithrombotic or thrombolytic therapy: American Society of Regional Anesthesia and Pain Medicine Evidence-Based Guidelines (Third Edition). Reg Anesth Pain Med. 2010 Jan-Feb;35(1):64-101. doi: 10.1097/aap.0b013e3181c15c70. PMID 20052816
- [Background] COVIDSurg Collaborative; GlobalSurg Collaborative. Timing of surgery following SARS-CoV-2 infection: an international prospective cohort study. Anaesthesia. 2021 Jun;76(6):748-758. doi: 10.1111/anae.15458. Epub 2021 Mar 9. PMID 33690889
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Bujang MA, Sa'at N, Sidik TMITAB, Joo LC. Sample Size Guidelines for Logistic Regression from Observational Studies with Large Population: Emphasis on the Accuracy Between Statistics and Parameters Based on Real Life Clinical Data. Malays J Med Sci. 2018 Jul;25(4):122-130. doi: 10.21315/mjms2018.25.4.12. Epub 2018 Aug 30. PMID 30914854
- [Derived] Nourouzpour N, Jen TTH, Bailey J, Jobin PG, Sutherland JM, Ho CM, Prabhakar C, Ke JXC. Association between anesthesia technique and death after hip fracture repair for patients with COVID-19. Can J Anaesth. 2024 Mar;71(3):367-377. doi: 10.1007/s12630-023-02673-2. Epub 2023 Dec 21. PMID 38129357

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT05133648/Prot_SAP_001.pdf